CLINICAL TRIAL: NCT06991751
Title: A Natural History of Cardiometabolic Disease Among US Bhutanese: Developing the Bhutanese Community of Central Ohio Health Study to Identify Synergizing Socioenvironmental and Biobehavioral Risk Factors Propagating Health Disparities From a Cross-Sectional Study
Brief Title: A Natural History of Cardiometabolic Disease Among US Bhutanese: Developing the Cross-Sectional Bhutanese Community of Central Ohio Health Study to Understand Acculturation as Synergizing Socioenvironmental and Biobehavioral Risk Factors Propagating ...
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002248; 002248-E
Record Dates: First submitted 2025-05-23; First posted 2025-05-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-29

CONDITIONS: Cardiometabolic Risk Factors; Mental Health
Keywords: Bhutanese; South Asian; Community engaged; Biospecimen perceptions; Epidemiology; Syndemic
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US Bhutanese: Those self-identifying as Bhutanese living in central Ohio.

SUMMARY:
Background:

As of 2021, almost 45 million people in the United States were foreign-born immigrants. South Asians, including people from Bhutan, are the fastest-growing immigrant subgroup in the US. Their income and education levels are higher than the US average. Yet they have worse physical and mental health outcomes than their White US-born counterparts. These risks include type 2 diabetes and obesity.

Objective:

This natural history study will explore how life experiences and environmental factors affect heart health and metabolism among Bhutanese people living in the US.

Eligibility:

Adults aged 18 years or older who identify as Bhutanese and live in the US.

Design:

Participants will be recruited and screened by the Bhutanese Community of Central Ohio (BCCO). They will have 1 visit to the BCCO s Arogya Clinic in Reynoldsburg. The visit will last 2 hours.

Participants will take a survey; they may use either English or Nepali. They will answer questions about their background; their experiences living in the US; and how their customs and habits might have changed. They will also be asked about their experiences with discrimination; their mental health and well-being; their community; quality of life; and overall physical health. The survey will take 60 minutes.

Participants will also speak with a researcher. They will be asked how they feel about providing biological samples; these may include saliva, blood, and urine. Their answers will be audio recorded.

DETAILED DESCRIPTION:
Study Description:

In 2021 we completed a cross-sectional feasibility study to assess cardiometabolic health of the Bhutanese refugee community in central Ohio. This is a cross-sectional pilot to assess the feasibility of establishing a long-term cohort study among the Bhutanese community to provide representation of a hardly-reached demographic group, optimize collection of behavioral and biological data. Schedule of Activities, describes the study activities including a survey assessing the participants experiences and a brief qualitative assessment examining the feasibility of obtaining biological samples.

Objectives:

The objectives are as follow:

Primary Objective: (Aim 1) To summarize socioecological characteristics of acculturation and cardiometabolic health from >=18-year-old adults United States Bhutanese living in Central Ohio.

Secondary Objectives: (Aim 2) To identify barriers and facilitators to biospecimen donation among United States Bhutanese adults living in Central Ohio.

Endpoints:

Primary Objective: (Aim 1) Summary on self-reported constructs of acculturation and acculturative stress, discrimination and stigma, health behaviors, medical history and health behaviors, mental health, sleep health, neighborhood social cohesion and community support, trauma, and medical history of cardiometabolic conditions.

Secondary Objectives: (Aim 2) Description of barriers and facilitators to biospecimen donation from US Bhutanese participants identified by qualitative inquiry and analysis of beliefs on biospecimens and invasiveness.

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in this study all of the following criteria must be met:

* Adults (aged 18 years and older) living in the United States
* Identify as Bhutanese, which will be defined as those individuals that resided or had/have their closest relatives residing in the Kingdom of Bhutan
* Bhutanese identity will also include those that self-identify as Bhutanese-Nepali or Bhutanese American

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any South Asian participants that do not identify as Bhutanese.
* Pregnant at time of study or screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older who identify as Bhutanese and live in the US, greater Ohio area.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To summarize socioecological characteristics of acculturation and cardiometabolic health from >=18-year-old adults United States Bhutanese living in Central Ohio. | 6-12 months
  Summary on self-reported constructs of acculturation and acculturative stress, discrimination and stigma, health behaviors, medical history and health behaviors, mental health, sleep health, neighborhood social cohesion and community support, trauma, and medical history of cardiometabolic conditions.

SECONDARY OUTCOMES:
To identify barriers and facilitators to biospecimen donation among United States Bhutanese adults living in Central Ohio. | 6-12 months
  Description of barriers and facilitators to biospecimen donation from US Bhutanese participants identified by qualitative inquiry and analysis of beliefs on biospecimens and invasiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra L Jackson, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Bhutanese Community of Central Ohio (BCCO), Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided